CLINICAL TRIAL: NCT00362726
Title: Effect of Atazanavir Administered With and Without Ritonavir on the Pharmacokinetics of the Cytochrome P450 2C8 Substrate Rosiglitazone in Healthy Subjects
Brief Title: Drug Interaction Study With Atazanavir Administered With and Without Ritonavir and a Cytochrome P450 Substrate Rosiglitazone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: AI424-106
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Rosiglitazone; Atazanavir Sulfate; Ritonavir

ARMS (5):
- A (Active Comparator)
  Interventions: Drug: Rosiglitazone maleate
- B (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate
- C (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate + Rosiglitazone maleate
- D (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate + Ritonavir
- E (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate + Ritonavir + Rosiglitazone maleate

INTERVENTIONS:
Drug: Rosiglitazone maleate — Tablets, Oral, RGZ 4 mg, once daily, 1 day.
  Arms: A
Drug: Atazanavir Sulphate — Capsules, Oral, ATV 400 mg, once daily, 5 days.
  Other Names: Reyataz
  Arms: B
Drug: Atazanavir Sulphate + Rosiglitazone maleate — Capsule, Oral, ATV 400 mg + RGZ 4 mg, once daily, 1 day.
  Other Names: Reyataz
  Arms: C
Drug: Atazanavir Sulphate + Ritonavir — Capsules, Oral, ATV 300 mg + RTV 100 mg, once daily, 14 days.
  Other Names: Reyataz
  Arms: D
Drug: Atazanavir Sulphate + Ritonavir + Rosiglitazone maleate — Capsules/Tablets, Oral, ATV 300 mg + RTV 100 mg + RGZ 4 mg, once daily, 1 day.
  Other Names: Reyataz
  Arms: E

SUMMARY:
The purpose of this clinical research study is to assess the effect of Atazanavir 400 mg QD and Atazanavir/Ritonavir 300/100 mg QD at steady state on the single dose pharmacokinetics of RGZ in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages 18 to 50 years old with a BMI 18 to 32 kg/m2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To assess the effect of Atazanavir 400 mg QD and Atazanavir/Ritonavir 300/100 mg QD at steady state on the single dose pharmacokinetics of Rosiglitazone in healthy subjects.

SECONDARY OUTCOMES:
To assess the safety and tolerability of Rosiglitazone and Atazanavir coadministration with and without Ritonavir.
To explore the relationship between Atazanavir exposure, CYP2C8 genotype and the pharmacokinetics of Rosiglitazone exposure

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hamilton, New Jersey, United States